CLINICAL TRIAL: NCT02135900
Title: The Use of Heliox in Obstructive Sleep Apnea Syndrome.
Acronym: HOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Michel Chalhoub, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-046
Record Dates: First submitted 2012-07-04; First posted 2014-05-12 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Heliox; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — heliox; Helium; Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heliox (Experimental): Heliox which is a mix of oxygen and helium gase will be administered through a face mask during part of the sleep study.
  Interventions: Drug: Heliox

INTERVENTIONS:
Drug: Heliox — From the onset of sleep until 2:00 am, patients will be placed on heliox 70/30. At 2:00 am patients will be switched to CPAP for titration according to American Academy of Sleep Medicine (AASM) guidelines.
  Other Names: Helium/Oxygen

SUMMARY:
The goals of the project is to evaluate the effects of Heliox therapy on obstructive sleep apnea syndrome (OSAS).

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common condition affecting up to 2-4 % of the general population. The pathophysiologic consequences of OSA include: excessive daytime sleepiness leading to increased car and work related accidents; and increased incidence of hypertension (HTN), stroke and possibly coronary artery events. In addition, patients with severe and untreated obstructive sleep apnea (OSA) have increased mortality compared to patients with treated severe OSA.The main stay of treatment of OSAS is the application of continuous positive airway pressure (CPAP) during sleep. The main problem with CPAP therapy is compliance. Heliox, a mixture of oxygen and helium has been used for many years in the treatment of upper airway obstruction. In this study, the investigators will evaluate the effectiveness of Heliox in the treatment of OSAS. Adult subjects with the diagnosis of obstructive sleep apnea syndrome who are referred for repeat sleep study for CPAP titration will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 or older with obstructive sleep apnea syndrome (OSAS) presenting for CPAP titration.

Exclusion Criteria:

* Professional singers.
* Television or Radio hosts.
* Disk Jockeys.
* Subjects requiring oxygen therapy.
* Subjects younger than 18 year old.
* Pregnant women.
* Patients with chronic obstructive pulmonary disease (COPD) with forced expiratory volume 1 (FEV1) less than 50%.
* History of anatomic upper airway obstruction.
* Uncontrolled asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Chalhoub, MD, Principal Investigator — Staten Island University Hospital
Locations (1):
- Sleep center, Staten Island University Hospital, Staten Island, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heliox
Started | 32 (32 subjects started the study. 50 subjects were screened.)
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Heliox
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index
Description: Assessment of Apnea/Hypopnea Index (AHI) at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Time Frame: Baseline and in 6-8 hours. The reported data are at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Population: Subjects with documented sleep apnea syndrome on nocturnal polysomnography
Measure: Mean (95% Confidence Interval); unit: Apneas or hypopneas per hour sleep
Arm/Group | Heliox
Number analyzed (Participants) | 30
Apneas or hypopneas per hour sleep
  At baseline ( without Heliox) | 42.71 [33.16 to 52.25]
  after 6-8 hours ( with Heliox) | 40.95 [32.68 to 49.23]

2. Primary Outcome: Apnea Index (AI)
Description: Assessment of Apnea Index (AI) at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Time Frame: Baseline and in 6-8 hours. The reported data are at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Population: Subjects with documented sleep apnea syndrome on nocturnal polysomnography
Measure: Mean (95% Confidence Interval); unit: Number of apneas per hour sleep
Arm/Group | Heliox
Number analyzed (Participants) | 30
Number of apneas per hour sleep
  At baseline ( without Heliox) | 16.46 [7.59 to 25.33]
  after 6-8 hours ( with Heliox) | 11.26 [4.98 to 17.53]

3. Primary Outcome: Lowest Oxygen Saturation (L SO2)
Description: Assessment of L SO2 at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Time Frame: Baseline and in 6-8 hours.
Population: Subjects with documented sleep apnea syndrome on nocturnal polysomnography
Measure: Mean (95% Confidence Interval); unit: Percentage of oxygen saturation
Arm/Group | Heliox
Number analyzed (Participants) | 30
Percentage of oxygen saturation
  At baseline ( without Heliox) | 84.22 [82.07 to 86.38]
  after 6-8 hours ( with Heliox) | 90.47 [88.71 to 92.23]

4. Primary Outcome: Mean Oxygen Saturation (M SO2)
Description: Assessment of M SO2 at baseline ( without heliox) and after 6-8 hours of sleep with heliox.
Time Frame: Baseline and in 6-8 hours.
Population: Subjects with documented sleep apnea syndrome on nocturnal polysomnography
Measure: Mean (95% Confidence Interval); unit: Percentage of oxygen saturation
Arm/Group | Heliox
Number analyzed (Participants) | 30
Percentage of oxygen saturation
  At baseline ( without Heliox) | 93.47 [92.50 to 94.43]
  after 6-8 hours ( with Heliox) | 96.29 [95.51 to 97.07]

ADVERSE EVENTS:
Arm/Group | Heliox
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes